CLINICAL TRIAL: NCT04057664
Title: Managing the Pain - a Group Therapy Based on the Bio-psycho-social Treatment Approach for Women With Chronic Pelvic Pain and Chronic Belly Pain
Brief Title: A Group Therapy Based on the Bio-psycho-social Treatment Approach for Women With Chronic Pelvic and Chronic Belly Pain
Status: Terminated | Type: Observational
Why Stopped: The group therapy program is no longer offered at the site, because other group therapies appear to be better integrated into patients' daily lives.
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2018-28
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pain, Chronic; Pain, Pelvic; Pain, Abdominal; Depression; Sex Disorder; Endometriosis
Keywords: Coping; Multidisciplinary; Group Therapy; Psychotherapy; Physiotherapy
MeSH Terms: conditions — Chronic Pain; Pelvic Pain; Abdominal Pain; Depression; Sexual Dysfunction, Physiological; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multidisciplinary Group Therapy: Multidisciplinary group therapy for women with chronic pelvic or belly pain
  Interventions: Behavioral: Learning of Coping Strategies

INTERVENTIONS:
Behavioral: Learning of Coping Strategies — Group sessions with psychotherapy and physiotherapy

SUMMARY:
The project investigates the situation of patients with chronic pelvic and chronic belly pain before and after our group therapy.

DETAILED DESCRIPTION:
To treat patients with chronic pelvic and belly pain in an interdisciplinary way, we developped a group therapy consisting of twelve sessions and a booster session. The therapy is based on the bio-psycho-social model of pain and includes group sessions of psychotherapy as well as physiotherapy.

All patients fill in questionnaires (concerning pain impact, pain chronicity, depression, anxiety, stress, well-being and sexuality) before and after the therapy as well as three and twelve months after.

ELIGIBILITY:
Inclusion Criteria:

Women with chronic pelvic pain or belly pain participating in our group therapy who give their consent to the analysis of their data for the study

Exclusion Criteria:

* No participation in the group therapy
* Finishing the group therapy prematurely (>3 missed sessions)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with chronic pelvic or belly pain, participating in our multimodal group therapy
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Pelvic Pain Impact Questionnaire (PPIQ) | baseline, 6 weeks, 3 months, 12 months
  Self reported questionnaire with 8 questions to assess the impact of pelvic pain on quality of life, daily activities and emotional life. Each questions is scored 0-4, yielding a total from 0 and 32.

SECONDARY OUTCOMES:
Change in Sexual Functioning Questionnaire (CSFQ-14) | baseline, 6 weeks, 3 months, 12 months
  Self-reported questionnaire with 14 questions assessing comorbidity- or medication-related sexual dysfunction. Each questions is scored using a 5-point Likert scale. Total scores range from 14 to 70, with lower scores indicating greater levels of sexual dysfunction.
Change in Female Sexual Distress Scale-Revised (FSDS-R) | baseline, 6 weeks, 3 months, 12 months
  Self-reported questionnaire assessing distress associated with sexual dysfunction. Each questions is scored using a 5-point Likert scale (0=never to 4=always). Total scores range from 0 to 52, with higher scores indicating greater levels of sexually related distress.
Change in Chronic Pain Grade Scale (CPGS) | baseline, 6 weeks, 3 months, 12 months
  Self-reported questionnaire with 3 questions assessing the presence of chronic pain at the site of injury. Each questions is scored using a 11-point Likert scale. Total scores range from 0 to 30, with higher scores indicating more pain.
Change in Depression | baseline, 6 weeks, 3 months, 12 months
  Subscale of Depression Anxiety and Stress Scale (DASS) questionnaire. Self-reported questionnaire with 14 questions assessing depression. Each questions is scored using a 4-point Likert scale (0=does not apply at all to 3=apply very much). Total sub-scores range from 0 to 42.
Change in Anxiety | baseline, 6 weeks, 3 months, 12 months
  Subscale of Depression Anxiety and Stress Scale (DASS) questionnaire. Self-reported questionnaire with 14 questions assessing anxiety. Each questions is scored using a 4-point Likert scale (0=does not apply at all to 3=apply very much). Total sub-scores range from 0 to 42.
Change in Stress | baseline, 6 weeks, 3 months, 12 months
  Subscale of Depression Anxiety and Stress Scale (DASS) questionnaire. Self-reported questionnaire with 14 questions assessing stress. Each questions is scored using a 4-point Likert scale (0=does not apply at all to 3=apply very much). Total sub-scores range from 0 to 42.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Pain Medicine, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No